CLINICAL TRIAL: NCT05263648
Title: Feasibility Study of Virtual Reality Software to Reduce Stress in Cancer Patients Receiving Radiation Therapy
Brief Title: Virtual Reality Software to Reduce Stress in Cancer Patients
Acronym: OU-SCC VR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to an issue with the software developer that cannot be resolved.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OU-SCC-Virtual Reality
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Head and Neck Cancer
Keywords: Virtual Reality; Radiation Therapy; Education; Distress; Stress
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Sessions (Other): Patients will undergo at least two VR sessions. One prior to and one during the course of radiation treatment.
  Interventions: Other: Virtual Reality Session

INTERVENTIONS:
Other: Virtual Reality Session — VR-based education sessions will be used to influence patients' perceived emotional and social distress while undergoing radiation therapy (RT).
  Emotional and social distress levels will be evaluated using questionnaires at baseline (prior to the first VR experience), at completion of RT, and at 30-60 days post RT.

SUMMARY:
The purpose of this study is to test the ability of virtual reality-based social support to increase patient adherence to radiation therapy by reducing patient distress.

DETAILED DESCRIPTION:
This study will involve patients who have been diagnosed with breast or head and neck cancer and are suitable to receive radiation therapy. It is a single arm pilot trial designed to provide information on the safety, feasibility, and impacts of incorporating virtual reality (VR) software into the treatment plan of patients receiving radiation therapy with the goal of increasing patient adherence to radiation therapy.

Patients will be provided with VR-based education sessions prior to and during the course of radiation therapy. Patients' emotional and social distress levels will be assessed with questionnaires to measure the impacts of the VR software. Patients will be in the study for up to 3 months during regular cancer care, but the total time for the study procedures is anticipated to be 2-4 hours in total. Results from this study will be for research only and will not impact treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Must be able to read and speak English
3. Diagnosis of breast or head and neck cancer
4. Treatment plan includes radiotherapy within the next 2 months
5. Signed study-specific informed consent prior to study entry

Exclusion Criteria:

1. Previous radiation therapy treatment
2. Neurologic deficits
3. Visual disorder
4. Neuro-psychiatric disorder
5. Use of neuro-psychiatric drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is accruing 10 males and 10 females (n=20) by self-identification. No other genders will be recruited.
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who complete 2 VR sessions | Up to 3 Months
  Percentage of patients who complete 2 VR sessions will be calculated.
Proportion of patients reporting ease of use for VR sessions | Up to 3 Months
  Patients will be given a survey on their VR sessions to measure the ease of use and ability to provide useful information.
Proportion of overall adherence to radiation therapy | Up to 3 Months
  Patient adherence to radiation treatment will be recorded and proportion of overall adherence will be calculated.

SECONDARY OUTCOMES:
Change in state trait anxiety scale | Up to 3 Months
  Change in state trait anxiety scale from baseline to follow-up will be calculated
Change in brief symptom inventory | Up to 3 Months
  Change in brief symptom inventory scale from baseline to follow-up will be calculated
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v2.0 - Social Isolation - Short Form 8a (SI) | Up to 3 Months
  Change in PROMIS Item Bank v2.0 - Social Isolation - Short Form 8a (SI) from baseline to follow-up will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Christina Henson, MD, Principal Investigator — Stephenson Cancer Center

IPD SHARING:
Plan to Share IPD: No